CLINICAL TRIAL: NCT02113709
Title: Determining the Efficacy of Full-time Occlusion Therapy in Severe Amblyopia at All Ages
Brief Title: Determining the Efficacy of Full-time Occlusion Therapy in Severe Amblyopia at Different Ages
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mughal Eye Trust Hospital (Other)
Responsible Party: Principal Investigator, Dr. Sameera Irfan, Consultant Ophthalmologist, Mughal Eye Trust Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIrfanMEHT
Record Dates: First submitted 2014-03-29; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Amblyopia; Strabismus
Keywords: Amblyopia; Strabismus; Occlusion therapy; Visual improvement
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Visual improvement (Experimental): To see how efficiently visual improvement occurs by Full-time Occlusion therapy with an eye patch in severe amblyopia.
  Interventions: Device: Occlusion therapy by Eye Patch; Device: Occlusion therapy

INTERVENTIONS:
Device: Occlusion therapy by Eye Patch — The good eye was occluded by a stick-on eye patch to stimulate the amblyopic eye and its neural connections to learn to see again.
Device: Occlusion therapy — To see how much improvement in visual acuity occurs by full-time occlusion therapy.
  Other Names: eye patch (commercially pre-packed)

SUMMARY:
Objective: To find out how much visual improvement is possible in severe amblyopia using full-time occlusion therapy with an eye patch and to see if improvement is influenced by the patient's age.

Methods: An interventional clinical trial of 115 consecutive cases with unilateral, severe amblyopia was conducted at a tertiary referral center from Jan 2010 to Oct 2012. Patients were divided into three age groups: 3-7 years (n= 38), 8-12 years (n=41), 13-35 years (n=36). After a complete ophthalmological examination by a single ophthalmologist, cases with organic visual loss were excluded; cases with previous part-time occlusion therapy that had failed were included in the study. Patients were given optimal refractive correction for a month, followed by full-time occlusion therapy along with near visual activities for 3-4 hours/day. The therapy was continued until maximum visual recovery was achieved (6/6 Snellen's). Therapy was gradually reduced and stopped. Patients were followed-up regularly for the next 18 months.

DETAILED DESCRIPTION:
Amblyopia, ('blunt vision' in Ancient Greek), also known as lazy eye, is a visual deficiency in an eye that is otherwise physically normal, or that is greater than would be expected from any structural abnormalities of the eye. There are unsubstantiated beliefs that it is more difficult to treat amblyopia in older age groups, that children that have already received failed amblyopia therapy do not respond to treatment and that full-time occlusion therapy may result in occlusion (disuse) amblyopia of the good eye. The aim of this study was to assess whether these beliefs are true. Materials and methods This was a prospective, interventional clinical trial of 115 consecutive cases with unilateral, severe amblyopia conducted at a tertiary referral center in Lahore, Pakistan, from January 2010 to October 2012. Eligibility criteria included an age of over three years, visual acuity in the amblyopic eye from 6/60 Snellen's or even counting fingers only, visual acuity in the sound eye of 6/6. A complete ophthalmic examination was performed by only one ophthalmologist (SI). This included examining the fixation pattern of both eyes, presence or absence of a phoria or a tropia by a cover-uncover test, fundus examination and color vision using Ishihara color plates. Any case with an organic cause for visual loss was excluded from the study after a thorough ophthalmological examination. Assessment of visual acuity of either eye for both near and distance acuity (Snellen's and ETDRS charts) refraction and Best Corrected Visual Acuity (BCVA) was performed by a trained optician who was masked to the study and patient's demographics.

ELIGIBILITY:
Inclusion Criteria:

* a visual acuity of 6/60 or 0.1-0.2 ETDRS in one eye and 6/6 or 1.0 ETDRS in the good eye
* strabismic amblyopia
* patients of any age were included.

Exclusion Criteria:

* structural damage to the eye (organic amblyopia)
* ametropic amblyopia

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity improvement | 3 months
  Full-time occlusion therapy of good eye was performed for 2-3 months while closely monitoring the vision of both the good and the amblyopic eye. Vision was assessed by EDTRS Charts as well as Snellen's Chart.

SECONDARY OUTCOMES:
improvement in stereopsis | 1 year
  as equal visual acuity is attained by both eyes, the stereopsis also improves. It was assessed by satandardized TNO plates with the patient wearing polarized glasses over their own corrective spectacles.

OTHER OUTCOMES:
Does the patched good eye develop occlusion amblyopia | 3 months
  The vision of patched good eye was meticulously monitored to note the development of occlusion amblyopia

CONTACTS AND LOCATIONS:
Overall Officials: Sameera Irfan, FRCS, Principal Investigator — Mughal Eye Trust Hospital, Lahore, Pakistan
Locations (1):
- Mughal Eye Trust Hospital, Lahore, Punjab Province, Pakistan